CLINICAL TRIAL: NCT00961649
Title: Safety and IOP-Lowering Efficacy of Brinzolamide/Brimonidine Fixed Combination Ophthalmic Suspension in Patients With Open-Angle Glaucoma and/or Ocular Hypertension
Brief Title: Safety and Efficacy of Brinzolamide/Brimonidine Fixed Combination
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-09-038
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension; Brinzolamide; Brimonidine; Intraocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brinz/Brim (Experimental): Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension and Vehicle: 1 drop each instilled in both eyes 3 times a day for 6 weeks. A time lapse of at least 10 minutes was required between instillations of each study drug.
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension; Other: Vehicle
- Brinz (Active Comparator): Brinzolamide ophthalmic suspension, 1% and Vehicle: 1 drop each instilled in both eyes 3 times a day for 6 weeks. A time lapse of at least 10 minutes was required between instillations of each study drug.
  Interventions: Drug: Brinzolamide ophthalmic suspension, 1%; Other: Vehicle
- Brim (Active Comparator): Brimonidine tartrate ophthalmic solution, 0.2% and Vehicle: 1 drop each instilled in both eyes 3 times a day for 6 weeks. A time lapse of at least 10 minutes was required between instillations of each study drug.
  Interventions: Drug: Brimonidine tartrate ophthalmic solution, 0.2%; Other: Vehicle
- Brinz+Brim (Active Comparator): Brinzolamide ophthalmic suspension, 1% and brimonidine tartrate ophthalmic solution, 0.2%: 1 drop each instilled in both eyes 3 times a day for 6 weeks. A time lapse of at least 10 minutes was required between instillations of each study drug.
  Interventions: Drug: Brinzolamide ophthalmic suspension, 1%; Drug: Brimonidine tartrate ophthalmic solution, 0.2%

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
  Arms: Brinz/Brim
Drug: Brinzolamide ophthalmic suspension, 1%
  Arms: Brinz; Brinz+Brim
Drug: Brimonidine tartrate ophthalmic solution, 0.2%
  Arms: Brim; Brinz+Brim
Other: Vehicle — Inactive ingredients used as placebo
  Arms: Brim; Brinz; Brinz/Brim

SUMMARY:
The purpose of this study was to compare the safety and intraocular pressure (IOP)-lowering efficacy of a new fixed combination of brinzolamide/brimonidine (Brinz/Brim) to:

* its individual components (Brinz and Brim), and
* the concomitant administration of Brinz and Brim (Brinz+Brim).

DETAILED DESCRIPTION:
This study consisted of 5 visits conducted during 2 sequential phases: the screening/eligibility phase, which included a screening visit and 2 eligibility visits, and the treatment phase, which included 2 on-therapy visits conducted at Week 2 and Week 6 (or early exit). A washout period based on previous ocular medication preceded Eligibility Visit 1. Subjects who met all inclusion/exclusion criteria at both eligibility visits were randomized to 1 of 4 study drug groups for 6 weeks. Study drug instillation began the morning after the second eligibility visit. The study was terminated by the sponsor out of caution due to microgel formation in the Brinz/Brim formulation. 13 remaining active subjects were discontinued. Further analysis revealed that neither the drop size nor the concentration of the active ingredients was affected.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Diagnosis of open-angle glaucoma or ocular hypertension, with mean intraocular pressure within protocol-specified range at eligibility visit/s.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential if pregnant, lactating, or not using highly effective birth control measures.
* Any form of glaucoma other than open-angle glaucoma.
* Severe central vision loss in either eye.
* Chronic, recurrent, or severe inflammatory eye disease.
* Ocular trauma within the preceding 6 months.
* Ocular infection or ocular inflammation within the preceding 3 months.
* Clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment.
* Best-corrected visual acuity score worse than 55 letters using the Early Treatment Diabetic Retinopathy Study chart.
* Other ocular pathology (including severe dry eye) that may, in the opinion of the Investigator, preclude the administration of study product.
* Ocular surgery within the preceding 6 months.
* Ocular laser surgery within the preceding 3 months.
* Any abnormality preventing reliable applanation tonometry.
* Any other conditions, including severe illness, which could make the patient, in the opinion of the Investigator, unsuitable for the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Teague, BS, Sr. Clinical Manager, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 investigational centers in the United States.
Pre-assignment Details: Of the 195 enrolled, 25 subjects did not meet inclusion/exclusion criteria and were exited from the study as screen failures prior to randomization. This reporting group includes all randomized subjects (170).
Groups:
- Brinz/Brim: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension and Vehicle: 1 drop each instilled in both eyes 3 times a day for 6 weeks
- Brinz+Brim: Brinzolamide ophthalmic suspension, 1% and brimonidine tartrate ophthalmic solution, 0.2%: 1 drop each instilled in both eyes 3 times a day for 6 weeks
- Brinz: Brinzolamide ophthalmic suspension, 1% and Vehicle: 1 drop each instilled in both eyes 3 times a day for 6 weeks
- Brim: Brimonidine tartrate ophthalmic solution, 0.2% and Vehicle: 1 drop each instilled in both eyes 3 times a day for 6 weeks
Period: Overall Study
Arm/Group | Brinz/Brim | Brinz+Brim | Brinz | Brim
Started | 41 | 44 | 44 | 41
Completed | 32 | 40 | 39 | 37
Not Completed | 9 | 4 | 5 | 4
Not completed — Adverse Event | 4 | 0 | 0 | 2
Not completed — Inadequate control of IOP | 0 | 0 | 0 | 1
Not completed — Patient has travel plans during holidays | 0 | 0 | 1 | 0
Not completed — Patient left to Mexico-family emergency | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 4 | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized subjects, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinz/Brim | Brinz+Brim | Brinz | Brim | Total
Number analyzed (Participants) | 41 | 44 | 44 | 41 | 170
Age, Customized [Number; unit: participants]
  18 to 64 years | 15 | 20 | 20 | 21 | 76
  ≥65 years | 26 | 24 | 24 | 20 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 26 | 25 | 96
  Male | 18 | 22 | 18 | 16 | 74
Region of Enrollment [Number; unit: participants]
  United States | 41 | 44 | 44 | 41 | 170

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intraocular Pressure (IOP) From Baseline to Each of the Assessment Time Points (8 AM, + 2 Hrs, + 7 Hrs, and + 9 Hrs) at Week 6 - Brinz/Brim, Brinz, Brim
Description: The study drug was instilled at 8 AM and +7 hours relative to the 8 AM dosing (approximately 15 minutes after conducting the IOP measurements). Intraocular pressure was measured by Goldmann applanation tonometry. One eye from each patient was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Intent-to-Treat (ITT) analysis data set was pre-specified for the comparison of Brinz/Brim to its individual components (Brinz and Brim).
Time Frame: Baseline, Week 6
Population: ITT: All subjects who received study drug and had at least 1 scheduled on-therapy study visit.
Measure: Least Squares Mean (Standard Error); unit: millimeters mercury (mmHg)
Arm/Group | Brinz/Brim | Brinz | Brim
Number analyzed (Participants) | 41 | 44 | 41
millimeters mercury (mmHg)
  Change from Baseline (BL) at 8 AM | -5.5 (0.51) | -5.7 (0.48) | -4.1 (0.50)
  Change from BL at +2 hours relative to 8 AM dosing | -8.5 (0.51) | -4.7 (0.48) | -5.3 (0.51)
  Change from BL at +7 hours relative to 8 AM dosing | -5.4 (0.51) | -2.8 (0.48) | -3.0 (0.51)
  Change from BL at +9 hours relative to 8 AM dosing | -6.8 (0.51) | -3.9 (0.48) | -5.9 (0.51)

2. Primary Outcome: Mean Change in Intraocular Pressure (IOP) From Baseline to Each of the Assessment Time Points (8 AM, +2 Hrs, +7 Hrs, and +9 Hrs) at Week 6 - Brinz/Brim, Brinz+Brim
Description: The study drug was instilled at 8 AM and +7 hours relative to the 8 AM dosing (approximately 15 minutes after conducting the IOP measurements). Intraocular pressure was measured by Goldmann applanation tonometry. One eye from each patient was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Per-Protocol (PP) analysis data set was pre-specified for the comparison of Brinz/Brim to Brinz+Brim.
Time Frame: Baseline, Week 6
Population: PP: All subjects who received study drug, satisfied inclusion/exclusion criteria, and had at least 1 scheduled on-therapy visit. Individual subject visits or data points were excluded if protocol criteria were violated at a subset of the subject's visits and the violations, in the opinion of the Medical Monitor, did not invalidate remaining visits.
Measure: Least Squares Mean (Standard Error); unit: millimeters mercury (mmHg)
Arm/Group | Brinz/Brim | Brinz+Brim
Number analyzed (Participants) | 38 | 41
millimeters mercury (mmHg)
  Change from Baseline (BL) at 8 AM | -5.5 (0.52) | -5.7 (0.50)
  Change from BL at +2 hours relative to 8 AM dosing | -8.4 (0.54) | -8.3 (0.52)
  Change from BL at +7 hours relative to 8 AM dosing | -5.0 (0.54) | -4.4 (0.52)
  Change from BL at +9 hours relative to 8 AM dosing | -6.3 (0.55) | -6.3 (0.53)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all subjects who were exposed to the study medications.
Description: An adverse event was defined as any untoward medical occurrence in a subject who was administered a study treatment regardless of whether or not the event had a causal relationship with the treatment. All AEs were obtained as solicited comments from the study subjects and as observations by the Investigator as outlined in the study protocol.
Arm/Group | Brinz/Brim | Brinz+Brim | Brinz | Brim
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/44 | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 10/41 | 8/44 | 9/44 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=41) | Brinz+Brim (N=44) | Brinz (N=44) | Brim (N=41)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Not related
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Not related
Chest pain (General disorders) | 0 | 1 | 0 | 0 — Not related
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=41) | Brinz+Brim (N=44) | Brinz (N=44) | Brim (N=41)
Vision blurred (Eye disorders) | 7 | 6 | 7 | 6
Ocular hyperaemia (Eye disorders) | 3 | 0 | 2 | 1
Eye pain (Eye disorders) | 0 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.